CLINICAL TRIAL: NCT02590627
Title: In-vivo Efficacy and Safety of Artemether/Lumefantrine Vs Dihydroartemisinin-piperaquine for Treatment of Uncomplicated Malaria and Assessment of Parasite Genetic Factors Associated With Parasite Clearance or Treatment Failure
Acronym: WB-Malaria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute for Medical Research, Tanzania (Other Government)
Collaborators: Ministry of Health and Social Welfare, Tanzania (Other Government); World Health Organization (Other)
Responsible Party: Principal Investigator, Dr. Geofrey Makenga, Research Scientist, National Institute for Medical Research, Tanzania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WB-Malaria- Tanzania.
Record Dates: First submitted 2014-07-13; First posted 2015-10-29 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Malaria
Keywords: Parasite clearance, Treatment failure
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Artemether-lumefantrine
  Interventions: Drug: Artemether-lumefantrine
- B (Experimental): Dihydroartemisinin-piperaquine
  Interventions: Drug: Dihydroartemisinin-piperaquine

INTERVENTIONS:
Drug: Artemether-lumefantrine — Artemether-lumefantrine
  Other Names: A
  Arms: A
Drug: Dihydroartemisinin-piperaquine — Dihydroartemisinin-piperaquine
  Other Names: B
  Arms: B

SUMMARY:
Drug efficacy testing is one of the most important tasks that is routinely undertaken by the National Malaria Control Program (NMCP) in Tanzania and has been recommended by the World health Organisation to monitor the efficacy of artemisinin based combination therapy (ACT) and possibly detect evolution/emergency of tolerance/resistance to these drugs. Currently, Artemether-lumefantrine (ALu) is the only ACT recommended by the Ministry of Health and Social Welfare and therefore testing of new ACTs such as dihydroartemisinin-piperaquine (DHA-PQ) is important because alternative drugs are urgently required. Meanwhile, NMCP is revising the guidelines for treatment of malaria in Tanzania and DHA-PQ has been earmarked as an alternative ACT to be used together with ALu. However, efficacy and safety data of DHA-PQ is missing since no studies have been done in Tanzania. Thus, a study is proposed to assess the efficacy and safety of DHA-PQ Vs ALu and provide important data which will enable the NMCP to make informed decisions; and possibly recommend DHA-PQ in the new Malaria treatment guidelines as the second line drug for the treatment of uncomplicated malaria in the country.

DETAILED DESCRIPTION:
Currently, Artemether-lumefantrine (ALu) is the only ACT recommended by the Ministry of Health and Social Welfare and therefore testing of new ACTs such as dihydroartemisinin-piperaquine (DHA-PQ) is important because alternative drugs are urgently required. Meanwhile, NMCP is revising the guidelines for treatment of malaria in Tanzania and DHA-PQ has been earmarked as an alternative ACT to be used together with ALu. However, efficacy and safety data of DHA-PQ is missing since no studies have been done in Tanzania. Thus, a study is proposed to assess the efficacy and safety of DHA-PQ Vs ALu and provide important data which will enable the NMCP to make informed decisions; and possibly recommend DHA-PQ in the new Malaria treatment guidelines as the second line drug for the treatment of uncomplicated malaria in the country.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 6 months - 10 years, without severe malnutrition and with a slide-confirmed mono-infection of P. falciparum, and asexual parasitemia between 250 - 200000 asexual parasites/µl will be included.
* Other inclusion criteria will include, absence of dangers signs (see Exclusion Criteria), axillary temperature > 37.5oC or a history of fever within the past 24 hours and ability to swallow oral medications.
* The ability and willingness to attend scheduled follow-up visits and an informed consent provided by parent or guardian will also be considered as important inclusion criteria without which a patient will not be enrolled into the study.
* Patients shall not be excluded on the basis of reported prior treatment with other anti-malarial drugs other than DHA-PQ within the past 24 hours if they have fever (axillary temperature > 37.50C) and parasitemia.
* Patients should have stable residence within the catchment area throughout the study period

Exclusion Criteria:

* The exclusion criteria will include: presence of general danger signs or signs of severe falciparum malaria according to the definitions of WHO (Appendix 6), severe anaemia (Hb < 5 g/dL) and mixed or mono-infection with species other the P. falciparum.
* Others will include severe malnutrition (defined as a child whose growth standard is below -3 z-score or symmetrical oedema involving at least one of the feet or a mid-upper arm circumference < 110 mm.
* Patients with febrile conditions due to diseases other than malaria (e.g. measles, acute lower respiratory tract infection, severe diarrhoea with dehydration) or other known underlying chronic or severe diseases (e.g. cardiac, renal and hepatic diseases and HIV/AIDS) will be excluded.
* Furthermore, patients under regular medication, which may interfere with anti-malarial pharmacokinetics and those with a history of hypersensitivity reactions or contraindications to the artemisinin-based therapy, piperaquine or the alternative treatment, will not be included into the study

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 509 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
parasitological cure on day 28 for ALu and 42 for DHA-PQ | 42 days
  non-adjusted and adjusted by PCR to account for new infections.

SECONDARY OUTCOMES:
parasite clearance after 72 hours. | 72 hours
  Microscope Blood slide for malaria reading 0 parasite.
parasitological cure on day 14 | 14 days
  Microscope Blood slide for malaria reading 0 parasite.
extended parasitological cure on day 42 for ALu and 63 for DHA-PQ | 63 days
  PCR and Microscope Blood slide for malaria parasitemia reading 0.
improvement in haemoglobin level at day 28 from the day 0 baseline | 28 days
reduction in gametocyte carriage at day 14 and day 28 from the day 0 baseline, | 28 days
occurrence and severity of adverse events and genomic profile of P.falciparum. | 63 days

CONTACTS AND LOCATIONS:
Overall Officials: Deus Ishengoma, PHD, Principal Investigator — National Institute for Medical Research; Celine Mandara, MD, Msc, Study Director — National Institute for Medical Research
Locations (2):
- Tanzania (2):
  - Ujiji Health Centre, Ujiji, Kigoma Region
  - Muheza Disignated District Hospital, Muheza, Tanga

REFERENCES:
- [Derived] Mandara CI, Kavishe RA, Gesase S, Mghamba J, Ngadaya E, Mmbuji P, Mkude S, Mandike R, Njau R, Mohamed A, Lemnge MM, Warsame M, Ishengoma DS. High efficacy of artemether-lumefantrine and dihydroartemisinin-piperaquine for the treatment of uncomplicated falciparum malaria in Muheza and Kigoma Districts, Tanzania. Malar J. 2018 Jul 11;17(1):261. doi: 10.1186/s12936-018-2409-z. PMID 29996849